CLINICAL TRIAL: NCT02338089
Title: Investigating the Effect of Pulsatile Administration of Oxytocin on the Desensitization of Human Myometrium In-vitro
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-06
Record Dates: First submitted 2015-01-09; First posted 2015-01-14 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-09

CONDITIONS: Postpartum Hemorrhage
Keywords: Uterine contraction; Oxytocin desensitization
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (no oxytocin) pretreatment (No Intervention): Physiological saline solution (PSS). Every 15-minutes, the PSS will be flushed and fresh PSS will be added.
- Continuous oxytocin (desensitizing) pretreatment (Active Comparator): Continuous oxytocin 10-5M. This desensitizing treatment is based on previous experiments in our laboratory demonstrating this phenomenon (reference 25 of Internal Review). The desensitizing pretreatment mimics the clinical setting of labor augmentation. Every 15-minutes, the 10-5M oxytocin will be flushed and fresh 10-5M oxytocin will be added.
  Interventions: Drug: Oxytocin
- Pulsatile oxytocin pretreatment (Active Comparator): 15-minutes of 10-5M oxytocin, followed by PSS for 15-minutes, followed by 10-5M oxytocin, followed by 15-minutes PSS, and so-on, for a total duration of two-hours,
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin — Oxytocin, 100 micromolar solution
  Other Names: pitocin
  Arms: Continuous oxytocin (desensitizing) pretreatment; Pulsatile oxytocin pretreatment

SUMMARY:
Postpartum hemorrhage (PPH) is a leading cause of maternal morbidity and mortality worldwide and is caused most commonly by poor uterine muscle (myometrium) tone after delivery. The first line agent used in the prevention and treatment of PPH is oxytocin.

Women who require augmentation of labor with intravenous oxytocin because of inadequate labor progression have been shown to be at increased risk of PPH. Typically, for augmentation of labor, oxytocin is used as a continuous infusion, with no consensus on the initial dose, its increments or maximal limit. High concentration continuous oxytocin infusions are not without theirs risks, which include hyperstimulation, fetal distress, as well as uterine rupture.

Studies have shown the clinical benefits of pulsatile oxytocin delivery for labor induction and augmentation with regards to requirement of less total oxytocin, similar uterine contractility and similar rates of caesarean delivery when used for labor induction and augmentation. However, the rate of PPH as a primary outcome measure has not been investigated. Therefore we currently do not know the effect of pulsatile oxytocin delivery on the rate of PPH.

The investigators hypothesize that the effect of myometrial desensitization following pulsatile oxytocin exposure would be lower when compared to continuous oxytocin exposure. These results will help in establishing whether myometrial contractility and sensitivity to oxytocin can be better preserved by delivery of pulsatile oxytocin, rather than continuous oxytocin for labor induction and augmentation, and thereby result in less PPH.

DETAILED DESCRIPTION:
Typically labor can be augmented by exposure to high levels of continuous oxytocin, for prolonged periods. The increased incidence of uterine atony and PPH following exogenous oxytocin administration during labor augmentation is related to myometrial oxytocin receptor desensitization to oxytocin.

Human clinical trials have shown the benefits of pulsatile oxytocin administration for labor induction and augmentation, which include requirement of less total oxytocin, similar uterine contractility and similar rates of cesarean delivery. However, the outcome of the effect on PPH is not currently known.

Characterization of the effect of pulsatile oxytocin on the desensitization of myometrium when compared to the effect of continuous oxytocin, may provide guidance for the delivery of pulsatile oxytocin for labor induction and augmentation to protect against the otherwise higher risk of PPH. Furthermore, the delivery of pulsatile oxytocin may be considered in subgroups who are already at higher risk of PPH, and require labor augmentation.

The investigators' previously validated in-vitro model provides a solid foundation for the study of myometrial contractility under controlled conditions, without any confounders that could be encountered in clinical settings.

The results of this study will provide insight into the level of desensitization of human myometrium following exposure to pulsatile oxytocin. Based on oxytocin dose-response curves after pretreatment to continuous oxytocin and pretreatment to pulsatile oxytocin, we will be able to determine the extent of desensitized myometrium following each delivery method.

ELIGIBILITY:
Inclusion Criteria:

* Patients who give written consent to participate in this study
* Patients with gestational age 37-41 weeks
* Non-laboring patients, not exposed to exogenous oxytocin
* Patients requiring primary Cesarean delivery or first repeat Cesarean delivery

Exclusion Criteria:

* Patients who refuse to give written informed consent
* Patients who require general anesthesia
* Patients who had previous uterine surgery or more than one previous Cesarean delivery
* Patients with any condition predisposing to uterine atony and postpartum hemorrhage, such as abnormal placentation, multiple gestation, preeclampsia, macrosomia, polyhydramnios, uterine fibroids, bleeding diathesis, chorioamnionitis, or a previous history of postpartum bleeding
* Emergency Cesarean section in labor
* Patients on medications that could affect myometrial contractility, such as nifedipine, labetolol or magnesium sulphate.

Ages: 16 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2015-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Motility Index | 8 hours
  Motility index (MI) takes into account both the amplitude and frequency of the myometrial contraction. It is a calculated outcome, based on the formula: frequency/(10 x amplitude).
  The analysis is undertaken by attaching myometrial strips between an isometric force transducer and the base of an organ bath chamber.

SECONDARY OUTCOMES:
Amplitude of contraction | 8 hours
  The maximum extent of uterine muscle contraction, measured in grams (g). The analysis is undertaken by attaching myometrial strips between an isometric force transducer and the base of an organ bath chamber.
Frequency of contraction | 8 hours
  The number of contractions in uterine muscle (myometrium) over 10 minutes, spontaneously and in response to an agonist.
  The analysis is undertaken by attaching myometrial strips between an isometric force transducer and the base of an organ bath chamber.
Integrated area under response curve (AUC) | 8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Mrinalini Balki, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Talati C, Carvalho JCA, Luca A, Balki M. The Effect of Intermittent Oxytocin Pretreatment on Oxytocin-Induced Contractility of Human Myometrium In Vitro. Anesth Analg. 2019 Apr;128(4):671-678. doi: 10.1213/ANE.0000000000002834. PMID 29401080